CLINICAL TRIAL: NCT04391127
Title: Efficacy and Safety of Hydroxychloroquine and Ivermectin in Hospitalized no Critical Patients Secondary to COVID-19 Infection: Randomized Controlled Trial
Brief Title: Hydroxychloroquine and Ivermectin for the Treatment of COVID-19 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A-09
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Two non-transparent bottles The first bottle will contain the initial treatment: Two ivermectin tablets, two hydroxychloroquine tablets, or two placebo tablets.
  The second bottle will contain the follow-up treatment (10 tablets): Two tablets will be indicated, which will be take 12 hours after ingestion of the initial bottle and then one tablet every 12 hours for 4 more days. This bottle will contain placebo and hydroxychloroquine according to the corresponding group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospitalized patients with COVID-19 QTc < 500 mseg (Experimental): Patients with confirmed COVID-19 infection by RT-qPCR SARS-CoV-2 or suspected by chest computed tomography with criteria of hospitalization because emergency medical criteria, with no need of critical care assistance. The risk of hydroxychloroquine complications will be assessed by QT corrected by Bazett formula. If QTc < 500 ms could be randomized to hydroxychloroquine, ivermectin or placebo.
  Interventions: Drug: Hydroxychloroquine; Drug: Ivermectin; Drug: Placebo
- Hospitalized patients with COVID-19 infection with QTc >500ms (Experimental): Patients with confirmed COVID-19 infection by RT-qPCR SARS-CoV-2 or suspected by chest computed tomography with criteria of hospitalization because emergency medical criteria, with no need of critical care assistance. The risk of hydroxychloroquine complications will be assessed by QT corrected by Bazett formula. If QTc > 500 ms could be randomized to ivermectin or placebo.
  Interventions: Drug: Ivermectin; Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine: 400 mg PO every 12 hours for one day. Subsequently 200 mg every 12 hours per 4 more days.
  Arms: Hospitalized patients with COVID-19 QTc < 500 mseg
Drug: Ivermectin — Ivermectin 12 mg PO every 24 hours for one day (in case of weight less than 80 kg) or 18 mg PO every 24 hours for one day (in case of weight over 80 kg) Subsequently this group will take two tablets of placebo 12 hrs after ivermectin ingestion and then one tablet of placebo each 12 hrs per 4 more days.
Drug: Placebo — Two tablets of placebo PO every 12 hours for one day. Subsequently one tablet of placebo every 12 hours per 4 more days.

SUMMARY:
Background: In December 2019, patients with pneumonia secondary to a new subtype of Coronavirus (COVID-19) were identified in China. In a few weeks the virus spread and cases started practically all over the world. In February 2020, the WHO declared a pandemic. Severe symptoms have been found in patients mainly with comorbidities and over 50 years of age. At this time there is no proven therapeutic alternative. In vitro studies and observational experiences showed that antimalarial drugs (Chloroquine and hydroxychloroquine) had antiviral activity and increased viral clearance. Ivermectin, on the other hand, has been shown in vitro to reduce viral replication and in an observational cohort, greater viral clearance with promising clinical results. So far there is no standard of treatment and clinical trials are needed to find effective treatment alternatives. Objective: To evaluate the safety and efficacy of treatment with hydroxychloroquine and ivermectin for serious COVID-19 infections in no critical hospitalized patients. Material and methods: Randomized controlled trial of patients diagnosed with respiratory infection by COVID-19, who present criteria for hospitalization. Randomization will be performed to receive hydroxychloroquine at a dose of 400 mg every 12 hours for one day and then 200 mg every 12 hours, to complete a 5-day treatment schedule. Group 2: Ivermectin 12 mg every 24 hours for one day (less than 80 kg) or Ivermectin 18 mg every 24 hours for one day (greater than 80 kg) + placebo until the fifth day. Group 3: Placebo. Prior to randomization, the risk of cardiovascular complications determined by corrected QT interval, related to hydroxychloroquine intake will be assessed. If the patient is at high risk, the allocation will be to ivermectin only or to placebo in an independent randomization, if the risk is low, any of the three groups could be assigned. Outcomes: The primary outcome will be discharge from hospital for improvement. The safety outcomes will be requirement of mechanical intubation, septic shock or death. Viral clearance will also be evaluated by means of PCR, which will be taken on the 5th day after admission, day 14 and 21.

DETAILED DESCRIPTION:
Background In late December 2019, the health authorities of the People's Republic of China reported several cases of pneumonia of unknown origin in Wuhan City, Hubei Province, China. On December 31, 2019, the Chinese Center for Disease Control and Prevention began etiological and epidemiological research on this disease. Three samples of bronchoalveolar lavage were taken from patients from the Jinyintan hospital in Wuhan and through various processes they came to identify a new coronavirus that they initially called on January 7, 2020 as: 2019-nCoV. On January 2020, the World Health Organization (WHO) made the first recommendations on the epidemiological surveillance of this new coronavirus.

On January 22, 2020, the first session of the Emergencies Committee was convened by WHO in Geneva, Switzerland and on January 30 Public Health Emergency of International Importance (ESPII) was declared to the 2019 outbreak.

On February 11, the International Committee on Virus Taxonomy made up of experts, based on the biology, species and type of virus isolated, names this new coronavirus as SARS-CoV-2 and responds to "Severe Acute Respiratory Syndrome Coronavirus 2 "(Severe Acute Respiratory Syndrome CoronaVirus 2 for its acronym in English), the WHO proposes that same day to call the disease caused by SARS-CoV-2 as COVID-19.

The first case reported in Latin America was in Brazil on February 26 and on the 28th of the same month, Mexico communicates its first confirmed case of the new coronavirus in a 35-year-old patient from a trip to Italy. Given the alarming levels of spread and severity of COVID-19, at a press conference on March 11, 2020, WHO Director-General Tedros Adhanom Ghebreyesus declares the SARS-CoV-2.5 outbreak as a pandemic.

IVERMECTIN The SARS-CoV-2 viral genome was rapidly sequenced to allow for a diagnostic test, epidemiological follow-up, and the development of preventive and therapeutic strategies, however, to date there is no evidence from clinical trials for any therapy that improves the evolution of patients suspected or confirmed with COVID-19.

New potential candidates for the treatment of this disease have emerged. A preclinical study showed that ivermectin, an FDA-approved antiparasitic drug, reduces the viral load of SARS-CoV-2 in vitro.

Ivermectin is a broad-spectrum antiparasitic that has shown antiviral activity against a broad group of viruses in recent years. It has been shown to inhibit the import of HIV viral integrase into the nucleus of human cells and also replication of the virus. It does something similar with other proteins of the SV40 virus and the dengue virus. It has also been shown to limit the infection of RNA viruses such as dengue, West Nile virus, Venezuelan equine encephalitis virus, and influenza virus. It has also been shown to be effective against DNA viruses such as pseudorabies of the mice. On the other hand, it has not been shown to be effective against the zika virus in mice, although this should be re-evaluated.

Studies on the SARS-CoV-1 coronavirus have revealed that the alpha/beta1 importin of the virus plays a role in infection in relation to intracellular signals of the capsid protein, which may have an impact on the division of host cells. Studies in cultures of infected cells show that ivermectin has a potent antiviral effect against SARS-CoV-2 and opens up hopeful expectations for using this antiparasitic in the early treatment of COVID-19 which is likely to help reduce the viral load, prevent progression to severe phase and limit person-to-person transmission. Therefore, the development of clinical protocols comparing it with other antivirals with alternate mechanisms of action is important and should be established as soon as possible.

In the study by Patel et al., Ivermectin was evaluated in a cohort of patients requiring invasive mechanical ventilation. In the ivermectin group, they were admitted to a dose of 150mcg/kg once they were intubated and observed a significant reduction in mortality, as well as significant reductions in the length of hospitalization and days in the intensive care unit.

Hydroxychloroquine Antimalarial drugs such as chloroquine (CQ) and hydroxychloroquine (HCQ) have been used for more than a century. They have been used not only for malaria but also in rheumatic conditions due to their anti-inflammatory properties and good safety profile. That is why, in the midst of a pandemic, the question of the use of antimalarials in the treatment and prophylaxis of covid-19 has been raised.

Kayaerts et al. demonstrated the inhibition of SARS-CoV by chloroquine in Vero E6 cells at different post-infection times. Vincent et al. demonstrated the dose-dependent inhibition effect of the virus on Vero E6 cells immediately after viral absorption and also 3 to 5 hours later. They also demonstrated that the cells pre-treated with CQ were refractory to the virus in addition to improving terminal glycosylation of the ACE2 receptor, decreasing the viral affinity for the receptor and also reducing the onset of infection. The above illustrates the possibility of using HCQ for prophylaxis or treatment against SARS-CoV. Due to the similarities of SARS-CoV-2 with the SARS virus, several studies have proposed the use of HCQ and CQ for management of the current pandemic.

Wang et al. tested the in vitro effect of several antivirals approved by the Food and Drug Administration (FDA) of the United States of America. Remdesivir showed blocking of viral infection after virus entry with an Effective Concentration of 50% (EC50) of 0.77 μM and a cytotoxic concentration of 50% (CC50) greater than 100μM. Chloroquine had an EC50 = 1.13μM, and a CC50 greater than 100μM and an EC90 of 6.9μM. Chloroquine was effective at the viral entry and post-entry level, while remdesivir was only effective at the post-entry level. The above suggests a possible use of CQ as a prophylactic for SARS-CoV-2.19 infection.

Yao et al. Also tested the effect of HCQ and CQ in vitro. They tested the pharmacological activity of chloroquine and hydroxychloroquine using Vero cells infected with SARS-CoV-2. Physiology-based pharmacokinetic models (PBPK) were implemented for both drugs separately integrating their in vitro data. Using PBPK models, hydroxychloroquine concentrations in the lung fluid were simulated under 5 different dosing regimens to explore the most effective regimen while considering the safety profile of the drug. In this study, it was found that HCQ (EC50 = 0.72 μM) is more potent than chloroquine (EC50 = 5.47 μM) in vitro. Based on the results of the PBPK models, a loading dose of 400 mg twice daily of orally administered hydroxychloroquine sulfate is recommended, followed by a maintenance dose of 200 mg twice daily for 4 days for infection by SARS-CoV-2, since it reached three times the potency of CQ phosphate when administered 500 mg twice a day 5 days in advance.

Gao et al. demonstrated the superiority of CQ over control treatment in more than 100 patients with respect to inhibition of exacerbation of pneumonia, improvement in lung imaging findings, promoting negative virus conversion and shortening the course of disease in more than 10 hospitals in China. Gautret et al. treated 20 patients with hydroxychloroquine and compared the results with 16 controls in France. They used PCR to measure viral load on days 3, 4, 5, and 6 post-inclusion. The treatment group had a higher mean age, but no gender difference was made between the two groups. Asymptomatic patients and patients with upper and lower respiratory tract infections were treated. They concluded that HCQ was effective in reducing viral load. The results on day 3 indicated that 50% of the patients treated with HCQ had a reduction in viral load (p = 0.005), on day 4 it showed a 60% reduction (p = 0.04) on day 5, a 65% reduction (p= 0.006) and on day 6, 70% of the patients showed a reduction in the viral load (p= 0.001). Furthermore, they described the synergistic effect of azithromycin when used in conjunction with HCQ to decrease viral load. Dual treatment showed a 100% decrease in viral load (p <0.001) for day 6, while hydroxychloroquine alone showed a 70% decrease.

In the recently published recommendations of the American Society for Infectious Diseases (IDSA) on April 11, 2020, it is established that in hospitalized patients with COVID-19, the use of HCQ / CQ should only be given in the context of a clinical trial.

The best evidence currently available has failed to demonstrate or exclude a beneficial effect of HCQ on the clinical progression of COVID-19, as inferred by radiological findings, or on viral clearance by means of PCR tests, although a somewhat higher proportion in the HCQ group experienced clinical improvement (RR: 1.47; 95% CI 1.02 - 2.11, p=0.04). However, the certainty in the evidence was rated as very low mainly due to small sample sizes, co-interventions, and risk of bias due to methodological limitations. Furthermore, the selected results should be considered indirect, since significant patient outcomes (eg, mortality, rate of progression to ARDS, and need for mechanical ventilation) were not available.

Studies evaluating the addition of azithromycin (AZ) to HCQ provided indirect comparisons of failure of virological clearance with historical controls. The observed risk of mortality among patients who received HCQ + AZ during the hospitalization was 3.4% (6/175 patients). However, an estimated mortality rate in an untreated cohort was not provided in the manuscript. Compared to the lack of viral clearance in historical controls (100% virological failure), 12 symptomatic patients were compared on day 5 or 6 of a separate hospital in France. Patients who received HCQ + AZ treatment experienced numerically fewer cases of virologic failure (43% combined virologic failure; 29/71 patients). There is very low certainty in this comparison of treatment effect, mainly due to very high risk selection bias, making any claims of effectiveness highly uncertain. Furthermore, relying on intermediate outcomes, such as viral clearance to determine important outcomes for the patient (including a reduction in the development of pneumonia, hospital or ICU admission, or the need for intubation) adds another layer of imprecision.

Finally, Barbosa et al conducted a comparative study of hospitalized adults with viral pneumonia secondary to SARS-CoV-2 during the last two weeks of March 2020. A group receiving HCQ and support measures against another group that only received support measures. The primary endpoints were the effect of hydroxychloroquine use on the need to increase respiratory support, change in lymphocyte count, and change in neutrophil-lymphocyte ratio. In this study, of 63 included patients, 32 were assigned to the HCQ arm. The administration of HCQ was associated with the need to increase the degree of ventilatory support compared to those who did not receive HCQ for 5 days (p = 0.013). The change in total lymphocytes in the HCQ group was not different from that in the group that only received support measures. These authors concluded that the use of HCQ tends to worsen the neutrophil / lymphocyte ratio compared to the group that only received supportive measures, in addition to the fact that the use of HCQ was found to increase the risk that the patient required ventilatory management with intubation.

Definition of the problem

Due to the high rate of spread of COVID-19 infection, associated with a high rate of hospitalization due to respiratory failure, empirical treatment of active agents in vitro has become a common practice.

Hydroxychloroquine and ivermectin have demonstrated viral inhibition in vitro and observational experiences have proposed them as potentially safe alternatives with clinical efficacy.

The proposed treatments have an adequate margin of safety, in addition to the fact that we have extensive clinical experience because they were previously used in humans to treat malaria, rheumatologic diseases, or parasitosis. Due to this, in conjunction with the urgent need to seek therapeutic alternatives, controlled studies are required without assuming efficacy.

Justification COVID-19 infection has collapsed health systems in industrialized countries due to the large number of patients requiring respiratory assistance. There is no standard treatment for the management of this infection and the focus has been on the already known life support and management of Adult Respiratory Failure Syndrome in critically ill patients. The treatments used empirically have an adequate safety profile due to the experience in other clinical settings. The use of these empirical alternatives should be based on clinical trials since efficacy and safety should not be assumed in the group of patients with COVID-19. The Miguel Hidalgo Centennial Hospital has been assigned as a hospitalization center for COVID-19 patients in Aguascalientes Mexico.

Hypothesis

Treatment with hydroxychloroquine or Ivermectin will be superior to placebo, with a shorter hospital stay and a lower rate of complications (intubation, septic shock, or death).

ELIGIBILITY:
Inclusion Criteria:

* RT-qPCR SARS-CoV-2 positivity or chest computed Tomography with suspected COVID-19 pneumonia
* Hospitalization by medical emergency staff criteria

Exclusion Criteria:

* Other confirmed viral active and acute infection

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Mean days of hospital stay | Three months
  Days from admission as a suspected case of COVID with hospitalization criteria until discharge
Rate of Respiratory deterioration, requirement of invasive mechanical ventilation or dead | Three months
  Respiratory deterioration defined by respiratory rate > 25 per minute, requirement of high oxygen supply (FiO2 > 80% ) to maintain oxygen saturation > 90 %, invasive mechanical ventilation or dead.
Mean of oxygenation index delta | Three months
  Daily delta of oxygenation index during the hospitalization

SECONDARY OUTCOMES:
Mean time to viral PCR negativization | 5, 14, 21 and 28 days after the first positive PCR
  Mean time to viral negativization of RT-qPCR SARS-CoV-2. Pre Specified time: 5, 14, 21 and 28 days after the first positive PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Manuel Arreola Guerra, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Lv DF, Ying QM, Weng YS, Shen CB, Chu JG, Kong JP, Sun DH, Gao X, Weng XB, Chen XQ. Dynamic change process of target genes by RT-PCR testing of SARS-Cov-2 during the course of a Coronavirus Disease 2019 patient. Clin Chim Acta. 2020 Jul;506:172-175. doi: 10.1016/j.cca.2020.03.032. Epub 2020 Mar 27. PMID 32229107
- [Background] Munster VJ, Koopmans M, van Doremalen N, van Riel D, de Wit E. A Novel Coronavirus Emerging in China - Key Questions for Impact Assessment. N Engl J Med. 2020 Feb 20;382(8):692-694. doi: 10.1056/NEJMp2000929. Epub 2020 Jan 24. No abstract available. PMID 31978293
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Gonzalez Canga A, Sahagun Prieto AM, Diez Liebana MJ, Fernandez Martinez N, Sierra Vega M, Garcia Vieitez JJ. The pharmacokinetics and interactions of ivermectin in humans--a mini-review. AAPS J. 2008;10(1):42-6. doi: 10.1208/s12248-007-9000-9. Epub 2008 Jan 25. PMID 18446504
- [Background] Boldescu V, Behnam MAM, Vasilakis N, Klein CD. Broad-spectrum agents for flaviviral infections: dengue, Zika and beyond. Nat Rev Drug Discov. 2017 Aug;16(8):565-586. doi: 10.1038/nrd.2017.33. Epub 2017 May 5. PMID 28473729
- [Background] Wagstaff KM, Sivakumaran H, Heaton SM, Harrich D, Jans DA. Ivermectin is a specific inhibitor of importin alpha/beta-mediated nuclear import able to inhibit replication of HIV-1 and dengue virus. Biochem J. 2012 May 1;443(3):851-6. doi: 10.1042/BJ20120150. PMID 22417684
- [Background] Yang SNY, Atkinson SC, Wang C, Lee A, Bogoyevitch MA, Borg NA, Jans DA. The broad spectrum antiviral ivermectin targets the host nuclear transport importin alpha/beta1 heterodimer. Antiviral Res. 2020 May;177:104760. doi: 10.1016/j.antiviral.2020.104760. Epub 2020 Mar 3. PMID 32135219
- [Background] Ketkar H, Yang L, Wormser GP, Wang P. Lack of efficacy of ivermectin for prevention of a lethal Zika virus infection in a murine system. Diagn Microbiol Infect Dis. 2019 Sep;95(1):38-40. doi: 10.1016/j.diagmicrobio.2019.03.012. Epub 2019 Mar 29. PMID 31097261
- [Background] Geleris J, Sun Y, Platt J, Zucker J, Baldwin M, Hripcsak G, Labella A, Manson DK, Kubin C, Barr RG, Sobieszczyk ME, Schluger NW. Observational Study of Hydroxychloroquine in Hospitalized Patients with Covid-19. N Engl J Med. 2020 Jun 18;382(25):2411-2418. doi: 10.1056/NEJMoa2012410. Epub 2020 May 7. PMID 32379955
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- See also: Statement on the second meeting of the International Health Regulations (2005) Emergency Committee regarding the outbreak of novel coronavirus 2019 (n-CoV) on 30 January 2020. — https://www.who.int/news-room/detail/30-01-2020-statement-on-the-second-meeting-of-the-international-health-regulations-(2005)-emergency-committee-regarding-the-outbreak-of-novel-coronavirus-(2019-ncov)
- See also: World Health Organization.Coronavirus disease (COVID-19) outbreak — http://www.who.int
- See also: Infectious Diseases Society of America. (I. D. America, Producer) Retrieved ABRIL de 2020 from IDSA Guidelines on the Treatment and Management of Patients with COVID-19 — http://www.idsociety.org/COVID19guidelines